CLINICAL TRIAL: NCT00404326
Title: A Phase II Study of Transcriptional Therapy With the DNA Demethylating Hydralazine and the HDAC Inhibitor Valproate Associated to Concomitant Cisplatin Chemoradiation in FIGO Stage III Cervical Cancer.
Brief Title: Hydralazine and Valproate Plus Cisplatin Chemoradiation in Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: National Council of Science and Technology, Mexico (Other); Psicofarma, S.A. De C.V. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005/013/ICI
Record Dates: First submitted 2006-11-25; First posted 2006-11-28 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-11

CONDITIONS: Cervical Cancer
Keywords: Cervical carcinoma; Epigenetic therapy; Hydralazine; Valproate; Microarray analysis
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Hydralazine; Valproic Acid

INTERVENTIONS:
Drug: Hydralazine and magnesium valproate
Procedure: Punch biopsy of the primary tumor

SUMMARY:
The current standard for locally advanced cervical cancer is concurrent cisplatin-based chemotherapy, however, the treatment results need to be improved. Epigenetic aberrations play an important role in cancer progression by silencing growth regulatory genes and there is now evidence that inhibitors of DNA methylation and HDAC inhibition synergize the radiation and chemotherapy effects.

Objective. To determine response rate, safety and biological effects of hydralazine and magnesium valproate when added to cisplatin chemoradiation.

Hypothesis. Hydralazine and magnesium valproate associated to chemoradiation will increase the clinical complete response rate to 95% as compared to 75% as seen in historical controls treated with cisplatin chemoradiation in FIGO stage IIIB patients.

Metodology. A total of 17 FIGO stage IIIB patients with histologically confirmed cervical carcinoma with no previous treatment will be included. Patients will be typed for acetylator status and and then receive either 182 or 83 mg of hydralazine, and magnesium valproate at 40mg/Kg from day -7 to the end of chemoradiation (external and brachytherapy). Clinical response rate, safety and transcriptome changes will be analyzed.

DETAILED DESCRIPTION:
Eligible patients after signing informed consent will undergo study evaluation and then typed for acetylator phenotype before receive either 182 or 83 mg of hydralazine, and magnesium valproate at 30mg/Kg from day -7 to the end of chemoradiation (external and brachytherapy. External beam radiation will be delivered by megavoltage equipment for a dose of 50gy (2Gy fraction from monday to friday) concurrently with cisplatin at 40mg/m2 for six weeks. Within one to two weeks, intracavitary brachytherapy (low-dose rate, Cesium sources) will be delivered to achieve at least 85Gy to point A. A punch biopsy from the primary tumor will be taken at entering the study and at day 8 of hydralazine and valproate treatment (before the first dose of cisplatin and radiation)to assess global gene expression profiling by microarray analysis. Blood samples will be taken to assess global DNA methylation, histone deacetylase activity and plasma levels of hydralazine and valproic acid.

Clinical response and toxicity will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* informed consent, histological diagnosis of cervical carcinoma (epidermoid, adenoesquamous and adenocarcinoma), clinical stage III B, untreated, aged 18-70 years, performance status 0-2 according to ECOG classification, and adequate liver, hematological and renal function, as defined by: hemoglobin >10 g/L, leukocytes >4000/mm3, platelets >100 000mm3; normal creatinine value and creatinine clearance >60 mL/min; total bilirubin < 1.5 upper normal limit value; no evidence of systemic disease or para-aortic lymph node involvement.

Exclusion Criteria:

* History of allergy to hydralazine or valproate; past or present condition of rheumatic disease, central nervous system disease, heart failure from aortic stenosis and postural hypotension as diagnosed by a physician; previous use of the experimental drugs (hydralazine and magnesium valproate) as well as if patients were pregnant or breast-feeding. Other exclusion criteria included uncontrolled systemic disease or infection.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-05; Study Completion 2006-11

PRIMARY OUTCOMES:
Clinical Response
Safety

SECONDARY OUTCOMES:
Gene expression profiling
Global DNA methylation
HDAC activity
Plasma levels hydralazine and valproic acid

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Duenas-Gonzalez, MD, PhD., Study Director — National Institute of Cancerologia, Mexico
Locations (1):
- National Institute of Cancerologia, Mexico City, TLALPAN, Mexico